CLINICAL TRIAL: NCT00831441
Title: Apixaban for Prevention of Acute Ischemic Events - 2 A Phase 3, Randomized, Double-Blind, Evaluation of the Safety and Efficacy of Apixaban In Subjects With a Recent Acute Coronary Syndrome
Brief Title: Phase III Acute Coronary Syndrome
Acronym: APPRAISE-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry); Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CV185-068; EUDRACT# 2008-008298-77
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2015-12

CONDITIONS: Acute Coronary Syndrome
Keywords: NOS
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — apixaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apixaban (Active Comparator)
  Interventions: Drug: Apixaban
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apixaban — Tablets, Oral, 5 mg, twice daily, until study end
  Other Names: BSM-562247
  Arms: Apixaban
Drug: Placebo — Tablets, Oral, 0 mg, twice daily, until study end
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if apixaban is superior to placebo for preventing cardiovascular death, non-fatal myocardial infarction, or ischemic stroke in subjects with a recent acute coronary syndrome

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome (ACS)
* Clinically stable
* Receiving standard of care for ACS

Exclusion Criteria:

* Severe hypertension
* Active bleeding or high risk for major bleeding
* Hemoglobin < 9 g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7484 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (785):
- United States (221):
  - Uab Medical Center, Birmingham, Alabama
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Heart Center Research, Llc, Huntsville, Alabama
  - North Phoenix Heart Center, Phoenix, Arizona
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - Nea Baptist Clinic, Jonesboro, Arkansas
  - Phase Care, Llc, Alameda, California
  - Cardiology Consultants Of Orange County, Anaheim, California
  - Beaver Medical Group, Banning, California
  - Local Institution, Chula Vista, California
  - Escondido Cardiology Associates, Inc., Escondido, California
  - William D. Bowden, D.O., Healdsburg, California
  - California Heart Specialists, Inc., Huntington Beach, California
  - Caring Clinical Research Corporation, Laguna Hills, California
  - Eisenstein, Isaac, Lakewood, California
  - Arvind J. Mehta, Md, Long Beach, California
  - Local Institution, Los Alamitos, California
  - Preciado Cardiology Incorporated, Los Angeles, California
  - East Bay Physicians Medical Group, Oakland, California
  - St. Joseph Heritage Medical Group, Orange, California
  - A.R.I. Clinical Trials, Inc., Redondo Beach, California
  - Coastal Multi-Specialty Research, Santa Ana, California
  - Radiant Research, Inc, Santa Rosa, California
  - Harbbor-Ucla Medical Center, Torrance, California
  - Rocky Mountain Cardiology, Boulder, Colorado
  - South Denver Cardiology Associates Pc, Littleton, Colorado
  - Drogue Medical, Llc, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Alfieri Cardiology, Newark, Delaware
  - Orlando Heart Specialists, Altamonte Springs, Florida
  - Palm Beach Heart Institute, Llc, Atlantis, Florida
  - Ronald L. Walsh, Do, Clearwater, Florida
  - The Heart And Vascular Institute Of Florida, Clearwater, Florida
  - Cardiovascular Specialist Of South Florida, Davie, Florida
  - David E. Perloff, Md, Fort Lauderdale, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Jacksonville Heart Center, Pa, Jacksonville, Florida
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - East Coast Institute For Research, Jacksonville, Florida
  - The Cardio Vascular Center P.A., Lake Mary, Florida
  - Alpha Medical Research, Llc, Melbourne, Florida
  - Melbourne Internal Medicine Associates (Mima), Melbourne, Florida
  - Glenn J. Barquet, Md, Miami, Florida
  - Miami Cardiology Clinical Research, L.L.C., Miami, Florida
  - Advanced Pharma Clinical Research, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Mediquest Research Group Inc., Ocala, Florida
  - Ocala Research Institute, Inc, Ocala, Florida
  - Florida Heart Group, Orlando, Florida
  - Orlando Heart Center, Orlando, Florida
  - Palm Beach Gardens Research Center Llc, Palm Beach Gardens, Florida
  - Local Institution, Pembroke Pines, Florida
  - Cardiology Consultants, Pensacola, Florida
  - Advent Clinical Research Centers, Inc., Pinellas Park, Florida
  - Cardio-Pulmonary Associates, Plantation, Florida
  - Avivo Clin Clinical Services, Port Orange, Florida
  - St. Augustine Cardiology Associates, Saint Augustine, Florida
  - Heartcare Research, Sarasota, Florida
  - Dr Kiran C Patel Research Institute At Pepin Heart Hospital, Tampa, Florida
  - Howard T. Tee, M.D., F.A.C.P., F.A.C.C., Vero Beach, Florida
  - Indian River Cardiovascular Associates, Inc, Vero Beach, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Cardiovascular Physicians Of North Atlanta, Atlanta, Georgia
  - Medical College Of Georgia, Augusta, Georgia
  - Columbus Cardiology Associates Pc, Columbus, Georgia
  - Georgia Heart Specialists, Covington, Georgia
  - Atlanta Institute For Medical Research, Inc, Decatur, Georgia
  - In-Quest Medical Research, Llc, Duluth, Georgia
  - Alta Pharmaceutical Research Center, Inc., Dunwoody, Georgia
  - North Georgia Medical Research, Ellijay, Georgia
  - Northeast Georgia Heart Cntr, Pc, Gainesville, Georgia
  - Mercer University School Of Medicine, Macon, Georgia
  - Well Star Cardiovascular Medicine, Pc, Marietta, Georgia
  - Southern Heart Research Institute, Llc, Riverdale, Georgia
  - Memorial Hospital Of Carbondale, Carbondale, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University Of Chicago Hospitals, Chicago, Illinois
  - Clinical Investigation Specialists, Inc, Gurnee, Illinois
  - Gateway Cardiology. P.C, Jerseyville, Illinois
  - Midwest Heart Foundation, Lombard, Illinois
  - Local Institution, Moline, Illinois
  - Illinois Heart & Lung Research, Normal, Illinois
  - Heartcare Midwest, Peoria, Illinois
  - Elkhart Clinic, Llc, Elkhart, Indiana
  - St Margaret Mercy Healthcare Centers, Hammond, Indiana
  - Krannertt Institute Of Cardiology, Indianapolis, Indiana
  - R. L.Roudebush Va Medical Center, Indianapolis, Indiana
  - The Care Group, Llc, Indianapolis, Indiana
  - Medical Consultants, Pc, Muncie, Indiana
  - Local Institution, Valparaiso, Indiana
  - Mcfarland Clinic Pc, Ames, Iowa
  - Iowa Heart Center, West Des Moines, Iowa
  - Midwest Cardiology Associates , P.C., Overland Park, Kansas
  - Kentucky Heart & Vascular Physicians, Ashland, Kentucky
  - Local Institution, Hazard, Kentucky
  - Cardiovascular Associates, Psc, Louisville, Kentucky
  - Research Integrity, Llc, Owensboro, Kentucky
  - Alexandria Cardiology Clinic, Alexandria, Louisiana
  - Clinical Research Network, Alexandria, Louisiana
  - Tulane University Hospital And Clinic, New Orleans, Louisiana
  - Overton Brooks V.A.M.C., Shreveport, Louisiana
  - Louisiana State University Health Sciences Center-Shreveport, Shreveport, Louisiana
  - Louisiana Heart Center, Slidell, Louisiana
  - Local Institution, Annapolis, Maryland
  - Delmarva Heart Research Foundation, Salisbury, Maryland
  - Peninsula Cardiology Associates, P.A., Salisbury, Maryland
  - Endeavor Medical Research, Plc, Alpena, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Local Institution, Detroit, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Thoracic And Cardiovascular Healthcare Foundation, Lansing, Michigan
  - Local Institution, Mount Pleasant, Michigan
  - Covenant Medical Center, Inc, Saginaw, Michigan
  - Great Lakes Heart & Vascular Institute, Pc, Saint Joseph, Michigan
  - William Beaumont Hospital-Troy, Troy, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Va Medical Center, Minneapolis, Minnesota
  - University Of Minnesota, Medical School, Minneapolis, Minnesota
  - St Cloud Hospital, Saint Cloud, Minnesota
  - University Of Mississippi Medical Center, Jackson, Mississippi
  - Local Institution, Jackson, Mississippi
  - Missouri Cardiovascular Specialists, Columbia, Missouri
  - Washington University School Of Medicine, St Louis, Missouri
  - Gateway Cardiology, P.C., St Louis, Missouri
  - Bryanlgh Heart Institute, Lincoln, Nebraska
  - Heart Consultants, Omaha, Nebraska
  - Alegent Health Clinic Heart & Vascular Specialists, Omaha, Nebraska
  - Local Institution, Brick, New Jersey
  - Central Jersey Medical Research Center, Elizabeth, New Jersey
  - Hamilton Cardiology Associates, Hamilton, New Jersey
  - Local Institution, Linden, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Central New Jersey Cardiology, South Plainfield, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Buffalo General Hospital, Buffalo, New York
  - Dr. Michael Sacher, Massapequa, New York
  - Hudson Valley Heart Center, Poughkeepsie, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - The University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina Heart Institute At East Carolina University, Greenville, North Carolina
  - Wake Med Heart Center, Raleigh, North Carolina
  - Wilmington Medical Research, Wilmington, North Carolina
  - Azalea Research Center, Wilmington, North Carolina
  - Local Institution, Fargo, North Dakota
  - Otfried N. Niedermaier, Md, Akron, Ohio
  - City Cardiology Associates, Barberton, Ohio
  - Cincinnati Veterans Affairs Medical Center, Cincinnati, Ohio
  - Fairfield Cardiac Cath Lab, Llc, Fairfield, Ohio
  - Genoa Medical Center, Genoa, Ohio
  - Middletown Cardiovascular Associates, Middletown, Ohio
  - Toledo Cardiology Consultants, Toledo, Ohio
  - Local Institution, Youngstown, Ohio
  - Cardiology Associates Of Southeastern Ohio, Zanesville, Ohio
  - Blue Stem Cardiology, Bartlesville, Oklahoma
  - Cor Clinical Research, Llc, Oklahoma City, Oklahoma
  - University Of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cardiovascular Associates, Oklahoma City, Oklahoma
  - St. Charles Health System, Inc., Bend, Oregon
  - Portland Preventive Cardiology, L.L.C., Portland, Oregon
  - Blair Medical Associates, Inc., Altoona, Pennsylvania
  - St. Lukes Cardiology Associates, Bethlehem, Pennsylvania
  - Consultants In Cardiovascular Diseases, Inc., Erie, Pennsylvania
  - Hamot Medical Center, Erie, Pennsylvania
  - Richard M. Kastelic M.D. & Associates, P.C., Johnstown, Pennsylvania
  - The Heart Group, Lancaster, Pennsylvania
  - Drexel University College Of Medicine, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania Cardiology Associates, Philadelphia, Pennsylvania
  - Va Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Pottstown Medical Specialists, Inc, Pottstown, Pennsylvania
  - Local Institution, Scranton, Pennsylvania
  - Buxmont Cardiology Associates, Pc, Sellersville, Pennsylvania
  - Moffit Heart & Vascular Group, Wormleysburg, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Anmed Health, Anderson, South Carolina
  - Carl Wilson Sofley, Jr., Md, Anderson, South Carolina
  - Lowcountry Medical Group, Beaufort, South Carolina
  - Columbia Cardiology, Columbia, South Carolina
  - Cardiology Assoicates, Pc/Black Hills Clinical Research Ctr, Rapid City, South Dakota
  - North Central Heart Institute, Sioux Falls, South Dakota
  - The Chattanooga Heart Institute, Chattanooga, Tennessee
  - The Stern Cardiovascular Center, Pa, Germantown, Tennessee
  - Research Associates Of Jackson, Jackson, Tennessee
  - Mountain State Health Alliance, Johnson City, Tennessee
  - Knoxville Heart Group, Knoxville, Tennessee
  - Access Clinical Trials, Nashville, Tennessee
  - Parkway Cardiology Associates, Pc, Oak Ridge, Tennessee
  - Amarillo Heart Clinical Research Institute Inc., Amarillo, Texas
  - Dallas Va Medical Center, Dallas, Texas
  - Cardiovascular Research Institute Of Dallas, Dallas, Texas
  - Heart Consultants Of North Texas, Dallas, Texas
  - Texas Health Research & Education Institute, Fort Worth, Texas
  - T&R Clinic, Fort Worth, Texas
  - Med Tech, Inc., Houston, Texas
  - Methodist Debakey Heart & Vascular Center, Houston, Texas
  - Centex Research, Pineloch Medical Clinic, Houston, Texas
  - Heart Care Center, Houston, Texas
  - Northwest Houston Cardiology, Pa, Houston, Texas
  - Texas Cardiac Center, Lubbock, Texas
  - Central Cardiovascular Institute Of San Antonio, San Antonio, Texas
  - Jose A. Perez, M.D., San Antonio, Texas
  - S.A.M. Clinical Research Center, San Antonio, Texas
  - Sugarland Cardiology Associates, Sugarland, Texas
  - Scott&White Memorial Hospital, Temple, Texas
  - Northwest Heart Center, Tomball, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - Utah Cardiology P.C, Layton, Utah
  - Bermisa Family Practice & Research Center, Chesapeake, Virginia
  - Zakhary, Bosh, Danville, Virginia
  - Heart Care Associates P.C., Hopewell, Virginia
  - The Cardiology Group Centra., Lynchburg, Virginia
  - Virginia Cardiolovascular Associates, Manassas, Virginia
  - Local Institution, Midlothian, Virginia
  - Sendara Cardiovasular Research Institute, Norfolk, Virginia
  - Virgina Commonwealth Universitymedical Center, Richmond, Virginia
  - Inland Cardiology Associates, Spokane, Washington
  - Franciscan Research Center, Tacoma, Washington
  - Dean And St. Mary'S Outpatient Center, Madison, Wisconsin
  - Wheaton Franciscan Healthcare St. Joseph, Milwaukee, Wisconsin
- Argentina (32):
  - Local Institution, Berazategui, Buenos Aires
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Local Institution, Ciudad Autonoma de Beunos Aire, Buenos Aires
  - Local Institution, Coronel Suárez, Buenos Aires
  - Local Institution, Gaba, Buenos Aires
  - Local Institution, Haedo, Buenos Aires
  - Local Institution, Junín, Buenos Aires
  - Local Institution, La Plata, Buenos Aires
  - Local Institution, Lanús Oeste, Buenos Aires
  - Local Institution, Morón, Buenos Aires
  - Local Institution, Quilmes, Buenos Aires
  - Local Institution, Ramos Mejía, Buenos Aires
  - Local Institution, San Isidro, Buenos Aires
  - Local Institution, San Martín, Buenos Aires
  - Local Institution, Resistencia, Chaco Province
  - Local Institution, Corrientes, Corrientes Province
  - Local Institution, Corrientes Capital, Corrientes Province
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Villa Cabrera, Córdoba Province
  - Local Institution, Villa Carlos Paz, Córdoba Province
  - Local Institution, Villa María, Córdoba Province
  - Local Institution, San Salvador de Jujuy, Jujuy Province
  - Local Institution, Capital, Mendoza Province
  - Local Institution, Posadas, Misiones Province
  - Local Institution, Cipolletti, Río Negro Province
  - Local Institution, Salta, Salta Province
  - Local Institution, San Luis, San Luis Province
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, Santa Fe, Santa Fe Province
  - Local Institution, San Miguel de Tucumán, Tucumán Province
- Australia (13):
  - Local Institution, Bruce, Australian Capital Territory
  - Local Institution, Broken Hill, New South Wales
  - Local Institution, Kogarah, New South Wales
  - Local Institution, Lismore, New South Wales
  - Local Institution, Cairns, Queensland
  - Local Institution, Herston, Queensland
  - Local Institution, Milton, Queensland
  - Local Institution, Ashford, South Australia
  - Local Institution, Elizabeth Vale, South Australia
  - Local Institution, Woodville, South Australia
  - Local Institution, Fitzroy, Victoria
  - Local Institution, Geelong, Victoria
  - Local Institution, Richmond, Victoria
- Austria (5):
  - Local Institution, Feldkirch
  - Local Institution, Graz
  - Local Institution, Linz
  - Local Institution, Oberpullendorf
  - Local Institution, Vienna
- Belgium (12):
  - Local Institution, Antwerp, Antwerpen
  - Local Institution, Aalst
  - Local Institution, Anderlecht
  - Local Institution, Bonheiden
  - Local Institution, Brasschaat
  - Local Institution, Bruges
  - Local Institution, Ghent
  - Local Institution, Huy
  - Local Institution, Ieper
  - Local Institution, Mechelen
  - Local Institution, Mol
  - Local Institution, Yvoir
- Brazil (27):
  - Local Institution, Maceió, Alagoas
  - Local Institution, Sobral, Ceará
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Brasília, Federal District
  - Local Institution, Goiânia, Goiás
  - Local Institution, Juiz de Fora, Mato Grosso
  - Local Institution, Belo Horizonte, Minas Gerais
  - Local Institution, Belo Horzonte, Minas Gerais
  - Local Institution, Uberlândia, Minas Gerais
  - Local Institution, Curitiba, Paraná
  - Local Institution, Londrina, Paraná
  - Local Institution, Belém, Pará
  - Local Institution, Recife, Pernambuco
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Rio Janeiro, Rio de Janeiro
  - Local Institution, Natal, Rio Grande do Norte
  - Local Institution, Passo Fundo, Rio Grande do Sul
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Blumenau, Santa Catarina
  - Local Institution, São José, Santa Catarina
  - Local Institution, Campinas, São Paulo
  - Local Institution, Limeira, São Paulo
  - Local Institution, Marília, São Paulo
  - Local Institution, Santo André, São Paulo
  - Local Institution, São Caetano do Sul, São Paulo
  - Local Institution, São José do Rio Preto, São Paulo
  - Local Institution, São Paulo, São Paulo
- Bulgaria (8):
  - Local Institution, Burgas
  - Local Institution, Dimitrovgrad
  - Local Institution, Pazardzhik
  - Local Institution, Pleven
  - Local Institution, Plovdiv
  - Local Institution, Sofia
  - Local Institution, Stara Zagora
  - Local Institution, Varna
- Canada (27):
  - Local Institution, Edmonton, Alberta
  - Local Institution, New Westminster, British Columbia
  - Local Institution, Penticton, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Sydney, Nova Scotia
  - Local Institution, Cambridge, Ontario
  - Local Institution, Greater Sudbury, Ontario
  - Local Institution, Grimsby, Ontario
  - Local Institution, Kitchener, Ontario
  - Local Institution, London, Ontario
  - Local Institution, Oshawa, Ontario
  - Local Institution, Parry Sound, Ontario
  - Local Institution, Sarnia, Ontario
  - Local Institution, Scarborough Village, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Windsor, Ontario
  - Local Institution, Chiccutimi, Quebec
  - Local Institution, Lévis, Quebec
  - Local Institution, Montreal, Quebec
  - Local Institution, Saint-Charles-Borromée, Quebec
  - Local Institution, Saint-Jérôme, Quebec
  - Local Institution, Sorel-Tracy, Quebec
  - Local Institution, St-Foy, Quebec
  - Local Institution, Terrebonne, Quebec
- Chile (8):
  - Local Institution, Osorno, Los Lagos Region
  - Local Institution, Punta Arenas, Magallanes Antartica
  - Local Institution, Temuco, Región de la Araucanía
  - Local Institution, Viña del Mar, Región de Valparaíso
  - Local Institution, Concepción, Región del Biobío
  - Local Institution, Talcahuano, Región del Biobío
  - Local Institution, Santiago, Santiago Metropolitan
  - Local Institution, Port Montt
- China (23):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Chongqing, Chongqing Municipality
  - Local Institution, Lanzhou, Gansu
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Nanning, Guangxi
  - Local Institution, Shijiazhuang, Hebei
  - Local Institution, Harbin, Heilongjiang
  - Local Institution, Wuhan, Hubei
  - Local Institution, Changsha, Hunan
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Suzhou, Jiangsu
  - Local Institution, Nanchang, Jiangxi
  - Local Institution, Changchun, Jilin
  - Local Institution, Dalian, Liaoning
  - Local Institution, Shenyang, Liaoning
  - Local Institution, Jinan, Shandong
  - Local Institution, Beijing, Shanghai Municipality
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Chengdu, Sichuan
  - Local Institution, Chongqing, Sichuan
  - Local Institution, Kunming, Yunnan
  - Local Institution, Hangzhou, Zhejiang
  - Local Institution, Xi'an
- Colombia (8):
  - Local Institution, Bogotá, Cundinamaral
  - Local Institution, Cartagena, Departamento de Bolívar
  - Local Institution, Cali, Valle del Cauca Department
  - Local Institution, Barranquilla
  - Local Institution, Bogotá
  - Local Institution, Floridablanca
  - Local Institution, Manizales
  - Local Institution, Medellín
- Czechia (9):
  - Local Institution, Brno
  - Local Institution, Hradec Králové
  - Local Institution, Liberec
  - Local Institution, Nový Jičín
  - Local Institution, Olomouc
  - Local Institution, Ostrava
  - Local Institution, Prague
  - Local Institution, Rakovník
  - Local Institution, Ústí nad Orlicí
- Denmark (10):
  - Local Institution, Arhus C
  - Local Institution, Copenhagen
  - Local Institution, Esbjerg
  - Local Institution, Haderslev
  - Local Institution, Hellerup
  - Local Institution, Hillerød
  - Local Institution, Hvidovre
  - Local Institution, Næstved
  - Local Institution, Silkeborg
  - Local Institution, Slagelse
- Finland (4):
  - Local Institution, Espoo
  - Local Institution, Helsinki
  - Local Institution, Rovaniemi
  - Local Institution, Tampere
- France (11):
  - Local Institution, Albi
  - Local Institution, Amiens
  - Local Institution, Avignon
  - Local Institution, Cholet
  - Local Institution, Lagny-sur-Marne
  - Local Institution, Langres
  - Local Institution, Montpellier
  - Local Institution, Paris
  - Local Institution, Pau Universite Cedex
  - Local Institution, Strasbourg
  - Local Institution, Toulouse
- Germany (26):
  - Local Institution, Bad Berka
  - Local Institution, Bad Nauheim
  - Local Institution, Berlin
  - Local Institution, Bernau
  - Local Institution, Bonn
  - Local Institution, Chemnitz
  - Local Institution, Coswig
  - Local Institution, Cottbus
  - Local Institution, Dachau
  - Local Institution, Essen
  - Local Institution, Flensburg
  - Local Institution, Halle
  - Local Institution, Hamburg
  - Local Institution, Hoyerswerda
  - Local Institution, Jena
  - Local Institution, Leverkusen
  - Local Institution, Limburg
  - Local Institution, Lübeck
  - Local Institution, Mainz
  - Local Institution, Münster
  - Local Institution, Neuss
  - Local Institution, Paderborn
  - Local Institution, Pirna
  - Local Institution, Regensburg
  - Local Institution, Rostock
  - Local Institution, Wesel
- Hungary (15):
  - Local Institution, Baja
  - Local Institution, Balatonfüred
  - Local Institution, Budapest
  - Local Institution, Budpest
  - Local Institution, Cegléd
  - Local Institution, Debrecen
  - Local Institution, Dunaújváros
  - Local Institution, Hódmezővásárhely
  - Local Institution, Kecskemét
  - Local Institution, Miskolc
  - Local Institution, Szekszárd
  - Local Institution, Szentes
  - Local Institution, Székesfehérvár
  - Local Institution, Szombathely
  - Local Institution, Zalaegerszeg
- India (21):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Vijayawada, Andhra Pradesh
  - Local Institution, Ahmedabad, Gujarat
  - Local Institution, Vadodara, Gujarat
  - Local Institution, Gurgaon, Haryana
  - Local Institution, Bangalore, Karnataka
  - Local Institution, Mysore, Karnataka
  - Local Institution, Shivamogga, Karnataka
  - Local Institution, Indore, Madhya Pradesh
  - Local Institution, Mumbai, Maharashtra
  - Local Institution, Nagpur, Maharashtra
  - Local Institution, Pune, Maharashtra
  - Local Institution, Jalandhar, Punjab
  - Local Institution, Jaipur, Rajasthan
  - Local Institution, Chennai, Tamil Nadu
  - Local Institution, Coimbatore, Tamil Nadu
  - Local Institution, Lucknow, Uttar Pradesh
  - Local Institution, Bikaner
  - Local Institution, Mangalore
  - Local Institution, New Delhi
  - Local Institution, Pune
- Israel (13):
  - Local Institution, Afula
  - Local Institution, Ashkelon
  - Local Institution, Hadera
  - Local Institution, Haifa
  - Local Institution, Jerusalem
  - Local Institution, Kfar Saba
  - Local Institution, Nahariya
  - Local Institution, Nazareth
  - Local Institution, Petah Tikva
  - Local Institution, Rehovot
  - Local Institution, Safed
  - Local Institution, Tel Aviv
  - Local Institution, Tiberias
- Italy (16):
  - Local Institution, Ascoli Piceno
  - Local Institution, Bergamo
  - Local Institution, Chieti
  - Local Institution, Foggia
  - Local Institution, Gravedona (Co)
  - Local Institution, Grosseto
  - Local Institution, Massa
  - Local Institution, Milan
  - Local Institution, Naples
  - Local Institution, Novara
  - Local Institution, Pavia
  - Local Institution, Perugia
  - Local Institution, Roma
  - Local Institution, San Daniele Del Friuli (Udine)
  - Local Institution, Saronno (Va)
  - Local Institution, Verona
- Japan (41):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Seto-Shi, Aichi-ken
  - Local Institution, Matsudo, Chiba
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Kasuga, Fukuoka
  - Local Institution, Kurume, Fukuoka
  - Local Institution, Gifu, Gifu
  - Local Institution, Ogaki-Shi, Gifu
  - Local Institution, Kure, Hiroshima
  - Local Institution, Obihiro, Hokkaido
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kasama, Ibaraki
  - Local Institution, Tsuchiura-Shi, Ibaraki
  - Local Institution, Tsukuba, Ibaraki
  - Local Institution, Kanazawa, Ishikawa-ken
  - Local Institution, Kanoya, Kagoshima-ken
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Yokohama Sakae-Ku, Kanagawa
  - Local Institution, Yokosuka, Kanagawa
  - Local Institution, Kochi, Kochi
  - Local Institution, Kumamoto, Kumamoto
  - Local Institution, Kyoto, Kyoto
  - Local Institution, Ueda, Nagano
  - Local Institution, Beppu, Oita Prefecture
  - Local Institution, Ōita, Oita Prefecture
  - Local Institution, Osaka, Osaka
  - Local Institution, Sakai, Osaka
  - Local Institution, Saga, Saga-ken
  - Local Institution, Ureshino, Saga-ken
  - Local Institution, Ageo, Saitama
  - Local Institution, Koshigaya, Saitama
  - Local Institution, Toda, Saitama
  - Local Institution, Komatsushimachō, Tokushima
  - Local Institution, Chiyoda-Ku, Tokyo
  - Local Institution, Chuo-Ku, Tokyo
  - Local Institution, Hachiōji, Tokyo
  - Local Institution, Meguro City, Tokyo
  - Local Institution, Meguro-Ku, Tokyo
  - Local Institution, Tokyo, Tokyo
  - Local Institution, Iwakuni, Yamaguchi
  - Local Institution, Ube, Yamaguchi
- Mexico (18):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Cabo San Lucas, Baja Californa Sur
  - Local Institution, Chihuahua City, Chihuahua
  - Local Institution, Monclova, Coahuila
  - Local Institution, Durango, Durango
  - Local Institution, Tijuana, Estado de Baja California
  - Local Institution, Acapulco de Juárez, Guerrero
  - Local Institution, Pachuca, Hidalgo
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Querétaro City, Querétaro
  - Local Institution, San Luis Potosí City, San Luis Potosí
  - Local Institution, Culiacán, Sinaloa
  - Local Institution, Metepec, State of Mexico
  - Local Institution, Tlalnepantla, State of Mexico
  - Local Institution, Veracruz, Veracruz
  - Local Institution, Xalapa, Veracruz
- Netherlands (19):
  - Local Institution, Alkmaar
  - Local Institution, Almere Stad
  - Local Institution, Amsterdam
  - Local Institution, Beverwijk
  - Local Institution, Boxmeer
  - Local Institution, Dirksland
  - Local Institution, Ede
  - Local Institution, Goes
  - Local Institution, Gouda
  - Local Institution, Heerlen
  - Local Institution, Hilversum
  - Local Institution, Maastrict
  - Local Institution, Meppel
  - Local Institution, Purmerend
  - Local Institution, Sneek
  - Local Institution, The Hague
  - Local Institution, Veldhoven
  - Local Institution, Weert
  - Local Institution, Zwolle
- New Zealand (5):
  - Local Institution, Auckland
  - Local Institution, Christchurch
  - Local Institution, Hastings
  - Local Institution, Nelson
  - Local Institution, Palmerston North
- Norway (10):
  - Local Institution, Bergen
  - Local Institution, Bodø
  - Local Institution, Drammen
  - Local Institution, Hamar
  - Local Institution, Kongsvinger
  - Local Institution, Kristiansund
  - Local Institution, Lillehammer
  - Local Institution, Oslo
  - Local Institution, Stavanger
  - Local Institution, Tynset
- Peru (6):
  - Local Institution, Cusco, Departamento de Cusco
  - Local Institution, Ica, Ica
  - Local Institution, Chiclayo, Lambayeque
  - Local Institution, Lima, Lima Province
  - Local Institution, Bellavista, Provincia Constitucional del Callao
  - Local Institution, Callao, Provincia Constitucional del Callao
- Poland (28):
  - Local Institution, Węgrów, Mazowiekie
  - Local Institution, Bialystok
  - Local Institution, Bydgoszcz
  - Local Institution, Bytom
  - Local Institution, Częstochowa
  - Local Institution, Elblag
  - Local Institution, Gdynia
  - Local Institution, Grodzisk Mazowiecki
  - Local Institution, Inowrocław
  - Local Institution, Kielce
  - Local Institution, Kościerzyna
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Lublin
  - Local Institution, Opole
  - Local Institution, Ostrowiec Świętokrzyski
  - Local Institution, Poznan
  - Local Institution, Płock
  - Local Institution, Radom
  - Local Institution, Rzeszów
  - Local Institution, Szczecin
  - Local Institution, Słupsk
  - Local Institution, Tarnów
  - Local Institution, Torun
  - Local Institution, Warsaw
  - Local Institution, Włocławek
  - Local Institution, Zabrze
  - Local Institution, Zielona Góra
- Puerto Rico (2):
  - Local Institution, Cidra
  - Local Institution, San Juan
- Romania (10):
  - Local Institution, Arad
  - Local Institution, Baia Mare
  - Local Institution, Brăila
  - Local Institution, Bucharest
  - Local Institution, Craiova
  - Local Institution, Oradea
  - Local Institution, Piteşti
  - Local Institution, Sibiu
  - Local Institution, Târgu Mureş
  - Local Institution, Timișoara
- Russia (25):
  - Local Institution, Barnaul
  - Local Institution, Chelyabinsk
  - Local Institution, Kaluga
  - Local Institution, Kazan'
  - Local Institution, Kemerovo
  - Local Institution, Krasnoyarsk
  - Local Institution, Moscow
  - Local Institution, Moscow Reg. Zhekeznodorozhniy
  - Local Institution, Nizhny Novgorod
  - Local Institution, Novosibirsk
  - Local Institution, Odintsovo
  - Local Institution, Penza
  - Local Institution, Perm
  - Local Institution, Rostov-on-Don
  - Local Institution, Ryazan
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov
  - Local Institution, Tomsk
  - Local Institution, Tver'
  - Local Institution, Tyumen
  - Local Institution, Vasilievsky Island
  - Local Institution, Voronezh
  - Local Institution, Yaroslavl
  - Local Institution, Yekaterinburg
  - Local Institution, Zhukovskiy
- Local Institution, Singapore, Singapore
- Slovakia (8):
  - Local Institution, Banská Bystrica
  - Local Institution, Bratislava
  - Local Institution, Košice
  - Local Institution, Kráľovský Chlmec
  - Local Institution, Liptovský Hrádok
  - Local Institution, Lučenec
  - Local Institution, Martin
  - Local Institution, Nitra
- South Africa (12):
  - Local Institution, Port Elizabeth, Eastern Cape
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Centurion, Gauteng
  - Local Institution, Wapadrand - Pretoria, Gauteng
  - Local Institution, Durban, KwaZulu-Natal
  - Local Institution, Umhlanga, KwaZulu-Natal
  - Local Institution, Bellville, Western Cape
  - Local Institution, Kuils River, Western Cape
  - Local Institution, Pinelands, Western Cape
  - Local Institution, Somerset West, Western Cape
  - Local Institution, Worcester, Western Cape
  - Local Institution, Johannesburg
- South Korea (13):
  - Local Institution, Wŏnju, Gangwon-do
  - Local Institution, Yangsan, Gyeongangnam-Do
  - Local Institution, Anyang-si, Gyeonggi-do
  - Local Institution, Guri-si, Gyeonggi-do
  - Local Institution, Jinju, Gyeongsangam-Do
  - Local Institution, Daegu
  - Local Institution, Goyang
  - Local Institution, Gwangju
  - Local Institution, Incheon
  - Local Institution, Jeonbuk
  - Local Institution, Pusan
  - Local Institution, Seoul
  - Local Institution, Suwon
- Spain (21):
  - Local Institution, Villajoyosa, Alicante
  - Local Institution, Almería, Almeria
  - Local Institution, Oviedo, Asturas
  - Local Institution, Cáceres, Caceres
  - Local Institution, Figueres, Gerona
  - Local Institution, Madrid, Madrid
  - Local Institution, San Sebastián de los Reyes, Madrid
  - Local Institution, Santiago de Compostela, Santiago de Compostela
  - Local Institution, Barcelona
  - Local Institution, El Ejido
  - Local Institution, Granada
  - Local Institution, Lleida
  - Local Institution, Lugo
  - Local Institution, Madrid
  - Local Institution, Málaga
  - Local Institution, Seville
  - Local Institution, Tarragona
  - Local Institution, Torrevieja
  - Local Institution, Valencia
  - Local Institution, Valladolid
  - Local Institution, Zaragoza
- Sweden (12):
  - Local Institution, Eskilstuna
  - Local Institution, Halmstad
  - Local Institution, Helsingborg
  - Local Institution, Karlskoga
  - Local Institution, Karlstad
  - Local Institution, Köping
  - Local Institution, Lidköping
  - Local Institution, Mölndal
  - Local Institution, Skövde
  - Local Institution, Stockholm
  - Local Institution, Uppsala
  - Local Institution, Vaxjo
- Switzerland (4):
  - Local Institution, Lugano, Canton Ticino
  - Local Institution, Geneva
  - Local Institution, Sankt Gallen
  - Local Institution, Zurich
- Turkey (Türkiye) (8):
  - Local Institution, Beşevler, Ankara
  - Local Institution, Isanbul, Haseki
  - Local Institution, Bornova, İzmir
  - Local Institution, Ankara
  - Local Institution, Diyarbakır
  - Local Institution, Isparta
  - Local Institution, Konya
  - Local Institution, Kırıkkale
- Ukraine (14):
  - Local Institution, Chernivtsy
  - Local Institution, Dnipropetrovsk
  - Local Institution, Donetsk
  - Local Institution, Ivano-Frankivsk
  - Local Institution, Kharkiv
  - Local Institution, Kyiv
  - Local Institution, Luhansk
  - Local Institution, Lutsk
  - Local Institution, Lviv
  - Local Institution, Mykolayiv
  - Local Institution, Odesa
  - Local Institution, Simferopol
  - Local Institution, Vinnitsa
  - Local Institution, Zhaporizhzhya
- United Kingdom (19):
  - Local Institution, Belfast, Antrim
  - Local Institution, Belfast, Armagh
  - Local Institution, Portadown, Armagh
  - Local Institution, Ayr, Ayrshire
  - Local Institution, Kilmarnock, Ayrshire
  - Local Institution, Cambridge, Cambridgeshire
  - Local Institution, Chesterfield, Derbyshire
  - Local Institution, Dumfries, Dumfriesshire
  - Local Institution, Cottingham, East Yorkshire
  - Local Institution, Basildon, Essex
  - Local Institution, Chelmsford, Essex
  - Local Institution, Romford, Essex
  - Local Institution, Royal Tunbridge Wells, Kent
  - Local Institution, Blackpool, Lancashire
  - Local Institution, Scunthorpe, Lincolnshire
  - Local Institution, Harrow, Middlesex
  - Local Institution, Worksop, Nottinghamshire
  - Local Institution, Doncaster, South Yorkshire
  - Local Institution, New Castle Upon Tyne, Tyne and Wear

REFERENCES:
- [Derived] Sharma A, Hagstrom E, Wojdyla DM, Neely ML, Harrington RA, Wallentin L, Alexander JH, Goodman SG, Lopes RD; Apixaban for Prevention of Acute Ischemic Safety Events APPRAISE-2 Steering Committee and Investigators. Clinical consequences of bleeding among individuals with a recent acute coronary syndrome: Insights from the APPRAISE-2 trial. Am Heart J. 2019 Sep;215:106-113. doi: 10.1016/j.ahj.2019.05.004. Epub 2019 May 11. PMID 31310855
- [Derived] Inohara T, Pieper K, Wojdyla DM, Patel MR, Jones WS, Tricoci P, Mahaffey KW, James SK, Alexander JH, Lopes RD, Wallentin L, Ohman EM, Roe MT, Vemulapalli S. Incidence, timing, and type of first and recurrent ischemic events in patients with and without peripheral artery disease after an acute coronary syndrome. Am Heart J. 2018 Jul;201:25-32. doi: 10.1016/j.ahj.2018.03.013. Epub 2018 Mar 28. PMID 29910052
- [Derived] Sherwood MW, Lopes RD, Sun JL, Liaw D, Harrington RA, Wallentin L, Laskowitz DT, James SK, Goodman SG, Darius H, Lewis BS, Gibson CM, Pieper KS, Alexander JH. Apixaban following acute coronary syndromes in patients with prior stroke: Insights from the APPRAISE-2 trial. Am Heart J. 2018 Mar;197:1-8. doi: 10.1016/j.ahj.2017.09.020. Epub 2017 Oct 24. PMID 29447769
- [Derived] Guimaraes PO, Lopes RD, Stevens SR, Zimerman A, Wruck L, James SK, Haque G, Giraldez RRCV, Alexander JH, Alexander KP. Reporting Clinical End Points and Safety Events in an Acute Coronary Syndrome Trial: Results With Integrated Collection. J Am Heart Assoc. 2017 Apr 24;6(4):e005490. doi: 10.1161/JAHA.117.005490. PMID 28438739
- [Derived] Hess CN, James S, Lopes RD, Wojdyla DM, Neely ML, Liaw D, Hagstrom E, Bhatt DL, Husted S, Goodman SG, Lewis BS, Verheugt FWA, De Caterina R, Ogawa H, Wallentin L, Alexander JH. Apixaban Plus Mono Versus Dual Antiplatelet Therapy in Acute Coronary Syndromes: Insights From the APPRAISE-2 Trial. J Am Coll Cardiol. 2015 Aug 18;66(7):777-787. doi: 10.1016/j.jacc.2015.06.027. PMID 26271059
- [Derived] Khan R, Lopes RD, Neely ML, Stevens SR, Harrington RA, Diaz R, Cools F, Jansky P, Montalescot G, Atar D, Lopez-Sendon J, Flather M, Liaw D, Wallentin L, Alexander JH, Goodman SG; Apixaban for Prevention of Acute Ischemic Safety Events (APPRAISE)-2 Steering Committee and Investigators. Characterising and predicting bleeding in high-risk patients with an acute coronary syndrome. Heart. 2015 Sep;101(18):1475-84. doi: 10.1136/heartjnl-2014-307346. Epub 2015 Jun 24. PMID 26109589
- [Derived] Mahaffey KW, Hager R, Wojdyla D, White HD, Armstrong PW, Alexander JH, Tricoci P, Lopes RD, Ohman EM, Roe MT, Harrington RA, Wallentin L. Meta-analysis of intracranial hemorrhage in acute coronary syndromes: incidence, predictors, and clinical outcomes. J Am Heart Assoc. 2015 Jun 18;4(6):e001512. doi: 10.1161/JAHA.114.001512. PMID 26089177
- [Derived] Alexander JH, Lopes RD, James S, Kilaru R, He Y, Mohan P, Bhatt DL, Goodman S, Verheugt FW, Flather M, Huber K, Liaw D, Husted SE, Lopez-Sendon J, De Caterina R, Jansky P, Darius H, Vinereanu D, Cornel JH, Cools F, Atar D, Leiva-Pons JL, Keltai M, Ogawa H, Pais P, Parkhomenko A, Ruzyllo W, Diaz R, White H, Ruda M, Geraldes M, Lawrence J, Harrington RA, Wallentin L; APPRAISE-2 Investigators. Apixaban with antiplatelet therapy after acute coronary syndrome. N Engl J Med. 2011 Aug 25;365(8):699-708. doi: 10.1056/NEJMoa1105819. Epub 2011 Jul 24. PMID 21780946
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7484 participants enrolled and 7392 were randomized. Reasons for non-randomization: 2 Adverse event (AE), 18 withdrew consent, 1 lost to follow up, 3 administrative reason by sponsor, 2 deaths, 51 no longer met criteria, 15 other.
Groups:
- Placebo BID: Placebo: Tablets, Oral, 0 mg, twice daily. The Treatment Period was planned to be completed after at least 938 participants had a primary efficacy endpoint confirmed by adjudication. After 7392 participants had been randomized into the study, an independent Data Monitoring Committee recommended that the study be terminated early due to a clinically important increase in bleeding among participants randomized to apixaban which was not offset by meaningful reductions in ischemic events. The Study terminated in Year 2.
- Apixaban 5 mg BID: Apixaban: Tablets, Oral, 5 mg, twice daily. The Treatment Period was planned to be completed after at least 938 participants had a primary efficacy endpoint confirmed by adjudication. After 7392 participants had been randomized into the study, an independent Data Monitoring Committee recommended that the study be terminated early due to a clinically important increase in bleeding among participants randomized to apixaban which was not offset by meaningful reductions in ischemic events. The Study terminated in Year 2.
Period: Randomized
Arm/Group | Placebo BID | Apixaban 5 mg BID
Started | 3687 | 3705
Treated | 3643 | 3672
Completed | 0 | 0
Not Completed | 3687 | 3705
Not completed — Death | 82 | 81
Not completed — Adverse Event | 248 | 321
Not completed — Emergency procedure | 2 | 2
Not completed — Elective procedure | 26 | 25
Not completed — Physician Decision | 26 | 35
Not completed — No longer met criteria | 13 | 19
Not completed — Withdrawal by Subject | 178 | 212
Not completed — Lost to Follow-up | 26 | 35
Not completed — Administrative reason by sponsor | 2780 | 2671
Not completed — poor/non-compliance | 30 | 38
Not completed — non-specified | 276 | 266
Period: Follow Up (30 Days)
Arm/Group | Placebo BID | Apixaban 5 mg BID
Started | 3508 (3508 participants entered the follow up period.) | 3529 (3529 participants entered the follow up period.)
Completed | 3375 | 3355
Not Completed | 133 | 174
Not completed — Withdrawal by Subject | 41 | 34
Not completed — Lost to Follow-up | 13 | 27
Not completed — Death | 63 | 86
Not completed — non-specified | 16 | 26
Not completed — missing end of study status | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Placebo: Placebo: Tablets, Oral, 0 mg, twice daily.
- Apixaban 5 mg BID: Apixaban: Tablets, Oral, 5 mg, twice daily.
- Total: Total of all reporting groups
Arm/Group | Placebo | Apixaban 5 mg BID | Total
Number analyzed (Participants) | 3687 | 3705 | 7392
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (11.05) | 65.3 (10.89) | 65.4 (10.97)
Age, Customized [Number; unit: participants] — Less than (<); Greater than, equal to (≥).
  participants
    < 65 years | 1512 | 1526 | 3038
    ≥ 65 and < 75 years | 1420 | 1440 | 2860
    ≥ 75 years | 755 | 739 | 1494
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1169 | 1209 | 2378
  Male | 2518 | 2496 | 5014
Region of Enrollment [Number; unit: participants]
  Russian Federation | 540 | 542 | 1082
  Puerto Rico | 13 | 17 | 30
  Singapore | 11 | 14 | 25
  United States | 450 | 455 | 905
  Austria | 58 | 56 | 114
  Sweden | 50 | 55 | 105
  Netherlands | 45 | 52 | 97
  China | 36 | 39 | 75
  Poland | 176 | 177 | 353
  Korea, Republic of | 88 | 89 | 177
  Brazil | 125 | 125 | 250
  Slovakia | 30 | 29 | 59
  France | 22 | 18 | 40
  Bulgaria | 100 | 102 | 202
  Chile | 30 | 26 | 56
  Colombia | 45 | 43 | 88
  Argentina | 131 | 125 | 256
  Romania | 78 | 80 | 158
  Hungary | 121 | 120 | 241
  Japan | 91 | 95 | 186
  Ukraine | 128 | 130 | 258
  United Kingdom | 24 | 21 | 45
  Switzerland | 18 | 20 | 38
  India | 396 | 398 | 794
  Spain | 81 | 79 | 160
  New Zealand | 13 | 9 | 22
  Canada | 126 | 128 | 254
  Czech Republic | 54 | 54 | 108
  Turkey | 9 | 11 | 20
  Belgium | 47 | 50 | 97
  Norway | 26 | 25 | 51
  Finland | 4 | 3 | 7
  Denmark | 37 | 34 | 71
  Italy | 23 | 21 | 44
  South Africa | 66 | 67 | 133
  Mexico | 161 | 161 | 322
  Israel | 73 | 66 | 139
  Australia | 15 | 23 | 38
  Peru | 66 | 66 | 132
  Germany | 80 | 80 | 160
Antiplatelet Therapy [Number; unit: participants]
  Dual Antiplatelet Therapy | 2965 | 2968 | 5933
  Single Antiplatelet Therapy | 722 | 737 | 1459
ACS Index Event [Number; unit: participants] — Participants were enrolled in the study only after experiencing an acute coronary syndrome (post-ACS) and were categorized as having ST-segment elevation myocardial infarction (STEMI), non-STEMI, or unstable angina.
  participants
    STEMI | 1412 | 1426 | 2838
    non-STEMI | 1582 | 1581 | 3163
    Unstable angina | 693 | 698 | 1391

OUTCOME MEASURES:

1. Primary Outcome: Event Rate of Cardiovascular Death, Myocardial Infarction, or Ischemic Stroke During the Intended Treatment Period - Randomized Participants
Description: Event rate was percent of participants with an event of cardiovascular (CV) death, myocardial infarction (MI), or ischemic stroke (number of participants with event/number randomized) per 100 patient (100-pt) years. Study was terminated early and last patient, last visit was in Year 2. Only events confirmed by the adjudication committee were included in the analyses. CV death included deaths due to CV causes (eg, cardiogenic shock, heart failure, arrhythmia/sudden death, cardiac rupture, ischemic stroke, pulmonary embolism, venous/arterial thrombotic events) and other sudden deaths for which an alternative cause was not identified. Intended Treatment Period: the period that started on the day of randomization and ended at the efficacy cut-off date (cut-off date: the date all sites were informed that study drug should be discontinued for all participants, 18 November 2010).
Time Frame: Randomization (Day 1) to first event (CV death, MI, ischemic stroke), up to March 2011, approximately 2 years
Population: All randomized participants were analyzed.
Measure: Number; unit: percentage of participants/100-pt years
Groups:
- Apixaban 5 mg BID: Apixaban: Tablets, Oral, 5 mg, twice daily. Study was terminated in Year 2.
Arm/Group | Placebo | Apixaban 5 mg BID
Number analyzed (Participants) | 3687 | 3705
percentage of participants/100-pt years | 13.96 | 13.20
Statistical Analysis 1: Comparison: Placebo vs Apixaban 5 mg BID; A test of superiority at the one-sided α = 0.025 significance level for the primary efficacy outcome was performed; Test type: Superiority or Other; p = 0.5094, Cox proportional hazard models; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.80 to 1.11]

2. Secondary Outcome: Event Rate of Unstable Angina (UA) During the Intended Treatment Period - Randomized Participants
Description: Unstable Angina (UA) defined as worsening or recurrent severe or repetitive angina symptoms at rest lasting at least 10 minutes with at least 2 of the following: New and dynamic electrocardiogram (ECG) changes; angina symptoms leading to inpatient hospitalization; angina symptoms leading to an unplanned or urgent cardiac catheterization, with or without revascularization, that showed evidence of hemodynamically and clinically significant stenosis. Event rate was percent of participants with an event of unstable angina (number of participants with event/number randomized) per 100 patient (100-pt) years. Only events confirmed by the adjudication committee were included in the analyses. Intended Treatment Period: the period that started on the day of randomization and ended at the efficacy cut-off date (cut-off date: the date all sites were informed that study drug should be discontinued for all participants, 18 November 2010).
Time Frame: Randomization (Day 1) to first event of UA, up to March 2011, approximately 2 years
Population: All randomized participants were analyzed.
Measure: Number; unit: percentage of participants/100-pt years
Groups:
- Apixaban 5 mg BID: Apixaban: Tablets, Oral, 5 mg, twice daily. Study was terminated at Year 2.
Arm/Group | Placebo | Apixaban 5 mg BID
Number analyzed (Participants) | 3687 | 3705
percentage of participants/100-pt years | 4.21 | 3.95
Statistical Analysis 1: Comparison: Placebo vs Apixaban 5 mg BID; Test type: Superiority or Other; p = 0.6702, Cox proportional hazard models; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.70 to 1.26]

3. Secondary Outcome: Event Rate of Stroke During the Intended Treatment Period - Randomized Participants
Description: Event rate was percent of participants with an event of stroke (number of participants with event/number randomized) per 100 patient (100-pt) years. Only events confirmed by the adjudication committee were included in the analyses. Diagnosis of stroke required a new, non-traumatic, focal neurological deficit of sudden onset, lasting at least 24 hours that was not due to a readily identifiable non-vascular cause (ie, brain tumor). All strokes were classified as hemorrhagic (documentation on imaging (eg computed tomography scan or magnetic resonance imaging) of hemorrhage in the cerebral parenchyma, or a subdural or subarachnoid hemorrhage), non-hemorrhagic/ischemic stroke, ischemic stroke with hemorrhagic conversion, or type unknown. Intended Treatment Period: the period that started on the day of randomization (Day 1) and ended at the efficacy cut-off date (notification of study termination).
Time Frame: Randomization (Day 1) to first event (stroke), up to March 2011, approximately 2 years
Population: All randomized participants were analyzed.
Measure: Number; unit: percentage of participants/100-pt years
Arm/Group | Placebo | Apixaban 5 mg BID
Number analyzed (Participants) | 3687 | 3705
percentage of participants/100-pt years | 1.85 | 1.65
Statistical Analysis 1: Comparison: Placebo vs Apixaban 5 mg BID; Test type: Superiority or Other; p = 0.6311, Cox proportional hazard models; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.57 to 1.40]

4. Secondary Outcome: Event Rate of Myocardial Infarction (MI) During the Intended Treatment Period - Randomized Participants
Description: MI took into account whether the participant had a recent percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) surgery. Selected key criteria: Elevation of cardiac biomarkers (eg, Creatine Kinase MB fraction (CKMB), Troponin T, Troponin I) above the upper reference limit (URL) plus ischemic symptoms, ECG changes, or imaging evidence of new loss of viable myocardium or new regional wall motion abnormality; Death of CV etiology with new ST-segment elevation or left bundle branch block (LBBB) or fresh intracoronary thrombus by angiography or at autopsy occurring before biomarkers could be obtained or before their appearance in the blood; Following a PCI, elevation of cardiac biomarkers more than 3*URL; Following CABG surgery, elevation of cardiac biomarkers more than 5*URL; New, significant (≥0.04 s) Q waves in ≥2 contiguous leads; Pathologic findings of acute MI. Intended Treatment Period: Day of randomization (Day 1) to efficacy cut-off notice.
Time Frame: Randomization (Day 1) to first event (MI), up to March 2011, approximately 2 years
Population: All randomized participants were analyzed.
Measure: Number; unit: percentage of participants/100-pt years
Arm/Group | Placebo | Apixaban 5 mg BID
Number analyzed (Participants) | 3687 | 3705
percentage of participants/100-pt years | 9.20 | 8.59
Statistical Analysis 1: Comparison: Placebo vs Apixaban 5 mg BID; Test type: Superiority or Other; p = 0.5086, Cox proportional hazard models; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.76 to 1.14]

5. Secondary Outcome: Event Rate of Stent Thrombosis During the Intended Treatment Period - Randomized Participants
Description: Stent thrombosis: Definite stent thrombosis considered to have occurred by either angiographic or pathological confirmation; Probable stent thrombosis considered to have occurred in the following cases: any unexplained death within the first 30 days after stent implantation; irrespective of the time after the procedure, any MI that was related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause; Possible stent thrombosis considered to have occurred with any unexplained death from 30 days after intracoronary stenting until end of study (in Year 2). Event rate was percent of participants with an event of stent thrombosis (number with event/number randomized) per 100-pt years. Only events confirmed by the adjudication committee were included in the analyses. Intended Treatment Period: Day of randomization (Day 1) to efficacy cut-off notice of study termination.
Time Frame: Randomization (Day 1) to first event (stent thrombosis), up to March 2011, approximately 2 years
Population: All randomized participants were analyzed.
Measure: Number; unit: percentage of participants/100-pt years
Arm/Group | Placebo | Apixaban 5 mg BID
Number analyzed (Participants) | 3687 | 3705
percentage of participants/100-pt years | 2.21 | 1.61
Statistical Analysis 1: Comparison: Placebo vs Apixaban 5 mg BID; Test type: Superiority or Other; p = 0.1502, Cox proportional hazard models; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.47 to 1.12]

6. Secondary Outcome: Event Rate of Composite of Cardiovascular Death, Myocardial Infarction, Unstable Angina, or Ischemic Stroke During the Intended Treatment Period - Randomized Participants
Description: Event rate was percent of participants with an event of CV death, MI, unstable angina (UA), or ischemic stroke (number of participants with event/number randomized) per 100-pt years. Only events confirmed by the adjudication committee were included in the analyses. Each type of event was counted once per participant, but participants could have been counted in multiple categories. Intended Treatment Period: Day of randomization (Day 1) to efficacy cut-off date (notification of study termination).
Time Frame: Randomization (Day 1) to first event (CV death, MI, UA, Ischemic Stroke, up to March 2011, approximately 2 years
Population: All randomized participants were analyzed.
Measure: Number; unit: percentage of participants/100-pt years
Arm/Group | Placebo | Apixaban 5 mg BID
Number analyzed (Participants) | 3687 | 3705
percentage of participants/100-pt years | 17.95 | 16.92
Statistical Analysis 1: Comparison: Placebo vs Apixaban 5 mg BID; Test type: Superiority or Other; p = 0.4317, Cox proportional hazard models; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.82 to 1.09]

7. Secondary Outcome: Event Rate of Composite of Cardiovascular Death, Fatal Bleed, Myocardial Infarction, or Stroke During the Intended Treatment Period - Randomized Participants
Description: Event rate was percent of participants with an event of CV death, fatal bleed, MI, or stroke (number of participants with event/number randomized) per 100 patient (100-pt) years. Only events confirmed by the adjudication committee were included in the analyses. CV death included deaths due to CV causes; Diagnosis of stroke required a new, non-traumatic, focal neurological deficit of sudden onset, lasting at least 24 hours that was not due to a readily identifiable non-vascular cause; Fatal bleeding defined as bleeding that Adjudication Committee determined was the primary cause of death or contributed directly to death; MI took into account whether the participant had a recent PCI or CABG surgery. Intended Treatment Period: Day of randomization (Day 1) to efficacy cut-off date (notification of study termination).
Time Frame: Randomization (Day 1) to first event (CV death, Fatal Bleed, MI, or stroke), up to March 2011, approximately 2 years
Population: All randomized participants were analyzed.
Measure: Number; unit: percentage of participants/100-pt years
Arm/Group | Placebo | Apixaban 5 mg BID
Number analyzed (Participants) | 3687 | 3705
percentage of participants/100-pt years | 14.27 | 13.97
Statistical Analysis 1: Comparison: Placebo vs Apixaban 5 mg BID; Test type: Superiority or Other; p = 0.8015, Cox proportional hazard models; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.83 to 1.15]

8. Secondary Outcome: Event Rate of Composite of All-Cause Death, Myocardial Infarction, or Stroke During the Intended Treatment Period - Randomized Participants
Description: Cause of death was determined by the principal condition that caused the death, not the immediate mode of death.
  CV death: included deaths due to CV causes. Non-CV death: included non-CV deaths caused primarily by a malignancy, infection, bleeding, trauma, non-CV system organ failure, or non-CV surgery. Unknown: included deaths that were not attributable to one of the above categories of CV death or to a non-CV cause. MI accounted whether the participant had a recent PCI or CABG surgery. Diagnosis of stroke required a new, non-traumatic, focal neurological deficit of sudden onset, lasting at least 24 hours that was not due to a readily identifiable non-vascular cause. Only events confirmed by the adjudication committee were included in analyses. Intended Treatment Period: Day of randomization (Day 1) to efficacy cut-off date (notification of study termination).
Time Frame: Randomization (Day 1) to first event (All Cause Death, MI, or Stroke), up to March 2011, approximately 2 years
Population: All randomized participants were analyzed.
Measure: Number; unit: percentage of participants/100-pt years
Arm/Group | Placebo | Apixaban 5 mg BID
Number analyzed (Participants) | 3687 | 3705
percentage of participants/100-pt years | 15.65 | 15.48
Statistical Analysis 1: Comparison: Placebo vs Apixaban 5 mg BID; Test type: Superiority or Other; p = 0.8948, Cox proportional hazard models; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.85 to 1.15]

9. Primary Outcome: Event Rate of Confirmed Major Bleeding Using Thrombolysis in Myocardial Infarction (TIMI) Criteria During the Treatment Period - Treated Participants
Description: TIMI Major Bleed Criteria: Fatal bleeding, intracranial hemorrhage, and clinically overt bleeding with a hemoglobin (Hgb) drop of ≥ 5 grams per deciliter (g/dL), or ≥15% absolute decrease in hematocrit. To account for transfusions, Hgb measurements were adjusted for transfusions. A transfusion of 1 unit of blood was assumed to result in an increase by 1 g/dL in Hgb or 3% in hematocrit. Event rate was percent of participants with an event of Major Bleed as per TIMI (number of participants with event/number randomized) per 100 patient (100-pt) years. Only events confirmed by the adjudication committee were included in the analyses. Treatment Period=events with onset from first dose to last dose plus 2 days.
Time Frame: From first dose to first occurrence of event (TIMI major bleeding) during Treatment Period (first dose to last dose + 2 days), up to March 2011, approximately 2 years
Population: All participants who received at least one dose of blinded study drug and signed informed consent were analyzed.
Measure: Number; unit: percentage of participants/100-pt years
Arm/Group | Placebo | Apixaban 5 mg BID
Number analyzed (Participants) | 3643 | 3672
percentage of participants/100-pt years | 0.91 | 2.40
Statistical Analysis 1: Comparison: Placebo vs Apixaban 5 mg BID; A point estimate and two-sided 95% confidence interval (CI) for relative risk, as measured by the hazard ratio and a p-value for the test of equality of rates (HR = 1) was calculated; Test type: Superiority or Other; p = 0.0006, Cox Proportional Hazard model; Hazard Ratio (HR) = 2.59, 95% CI 2-sided [1.50 to 4.46]

10. Secondary Outcome: Event Rate of Confirmed Major Bleeding Using International Society on Thrombosis and Hemostasis (ISTH) Criteria During the Treatment Period - Treated Participants
Description: ISTH Criteria: Acute clinically overt bleeding defined as new onset, visible bleeding or signs or symptoms suggestive of bleeding confirmed by imaging techniques, which can detect the presence of blood (eg, ultrasound, CT, MRI). Major bleeding: acute clinically overt bleeding accompanied by one or more of the following: A decrease in Hgb of 2 g/dL or more over 24 hours; A transfusion of 2 or more units of packed red blood cells (RBCs); Bleeding that occurs in at least one of the following sites: intracranial, intraspinal, intraocular (within the corpus of the eye; thus, a conjunctival bleed is not an intraocular bleed), pericardial, intra-articular, intramuscular with compartment syndrome, retroperitoneal; Bleeding that was fatal. Bleeding events were adjudicated by the Adjudication Committee. Event rate was percent of participants with an event (number with event/number randomized) per 100-pt years. Treatment Period=events with onset from first dose to last dose plus 2 days.
Time Frame: From first dose to first occurrence of event (ISTH major bleed) during Treatment Period (first dose to last dose + 2 days), up to March 2011, approximately 2 years
Population: All participants who received at least one dose of blinded study drug and signed informed consent were analyzed.
Measure: Number; unit: percentage of participants/100-pt years
Arm/Group | Placebo | Apixaban 5 mg BID
Number analyzed (Participants) | 3643 | 3672
percentage of participants/100-pt years | 2.04 | 5.13
Statistical Analysis 1: Comparison: Placebo vs Apixaban 5 mg BID; Test type: Superiority or Other; p < 0.0001, Cox Proportional Hazard model; Hazard Ratio (HR) = 2.48, 95% CI 2-sided [1.72 to 3.58]

11. Secondary Outcome: Event Rate of Confirmed Major Bleeding or Clinically Relevant Non-Major Bleeding (CRNM) Using ISTH Criteria During the Treatment Period - Treated Participants
Description: ISTH Major bleed: acute clinically overt bleeding accompanied by one or more of the following: A decrease in Hgb of 2 g/dL or more over 24 hours; A transfusion of 2 or more units of packed RBCs; Bleeding that occurs in at least one of the following critical sites: intracranial, intraspinal, intraocular (within the corpus of the eye), pericardial, intra-articular, intramuscular with compartment syndrome, retroperitoneal; Bleeding that was fatal. CRNM: acute clinically overt bleeding that did not satisfy additional criteria required for the bleeding event to be defined as a major bleeding event and meets at least one of the following: Hospital admission for bleeding; Physician guided medical or surgical treatment for bleeding; Change in anti-thrombotic treatment (anticoagulant or antiplatelet) therapy. Bleeding events were adjudicated by the Adjudication Committee. Treatment Period=events with onset from first dose to last dose plus 2 days.
Time Frame: From first dose to first occurrence of event (ISTH major or CRNM bleed) during Treatment Period (first dose to last dose + 2 days), up to March 2011, approximately 2 years
Population: All participants who received at least one dose of blinded study drug and signed informed consent were analyzed.
Measure: Number; unit: percentage of participants/100-pt years
Arm/Group | Placebo | Apixaban 5 mg BID
Number analyzed (Participants) | 3643 | 3672
percentage of participants/100-pt years | 2.29 | 6.15
Statistical Analysis 1: Comparison: Placebo vs Apixaban 5 mg BID; Test type: Superiority or Other; p < 0.0001, Cox Proportional Hazard model; Hazard Ratio (HR) = 2.64, 95% CI 2-sided [1.87 to 3.72]

12. Secondary Outcome: Event Rate of All Bleeding Reported by the Investigator During the Treatment Period - Treated Participants
Description: Bleeding events were adjudicated by the Adjudication Committee and classified according to Thrombolysis in Myocardial Infarction (TIMI) major, minor, minimal, and International Society on Thrombosis and Hemostasis (ISTH) major and clinically relevant non-major bleeding (CRNM) criteria. The adjudicated results based on TIMI and ISTH classifications, and programmatically identified events (not adjudicated) according to Global Use of Strategies to Open Occluded Coronary Arteries (GUSTO) classification were used in the analyses of bleeding endpoints. GUSTO Bleed Criteria included Severe or life-threatening: Intracranial hemorrhage, or bleeding that causes hemodynamic compromise requiring intervention; Moderate: Bleeding that requires a blood transfusion, but does not result in hemodynamic compromise; Mild: Bleeding that does not meet criteria for either severe or moderate bleeding. Treatment Period=events with onset from first dose to last dose plus 2 days.
Time Frame: From first dose to first occurrence of event (Bleeding) during Treatment Period (first dose to last dose + 2 days), up to March 2011, approximately 2 years
Population: All participants who received at least one dose of blinded study drug and signed informed consent were analyzed.
Measure: Number; unit: percentage of participants/100-pt years
Arm/Group | Placebo | Apixaban 5 mg BID
Number analyzed (Participants) | 3643 | 3672
percentage of participants/100-pt years | 16.33 | 39.98
Statistical Analysis 1: Comparison: Placebo vs Apixaban 5 mg BID; Test type: Superiority or Other; p < 0.0001, Cox Proportional Hazard model; Hazard Ratio (HR) = 2.36, 95% CI 2-sided [2.06 to 2.70]

ADVERSE EVENTS:
Arm/Group | Apixaban 5 mg BID | Placebo BID
Serious Adverse Events (participants affected / at risk) | 894/3672 | 884/3643
Other Adverse Events (participants affected / at risk) | 357/3672 | 231/3643
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban 5 mg BID (N=3672) | Placebo BID (N=3643)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Arteriospasm coronary (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 2 | 2
Bacterial tracheitis (Infections and infestations) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 6 | 3
Cardiac failure congestive (Cardiac disorders) | 16 | 17
Cardiomyopathy (Cardiac disorders) | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 20 | 39
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 5
Electrocardiogram QRS complex prolonged (Investigations) | 1 | 0
Embolism arterial (Vascular disorders) | 0 | 2
Erysipelas (Infections and infestations) | 0 | 1
Extravasation blood (Vascular disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 4
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 1
General physical health deterioration (General disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hepatic enzyme increased (Investigations) | 2 | 2
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 3 | 3
Hypertension (Vascular disorders) | 16 | 13
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Interventricular septum rupture (Cardiac disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Mediastinitis (Infections and infestations) | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Peripheral ischaemia (Vascular disorders) | 3 | 1
Pneumonia (Infections and infestations) | 35 | 35
Pneumonia bacterial (Infections and infestations) | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Sarcoidosis (Immune system disorders) | 2 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0
Sudden death (General disorders) | 19 | 13
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 5 | 6
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Vasospasm (Vascular disorders) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Anaphylactic shock (Immune system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 37 | 41
Aortic dissection (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 1
Arteriosclerosis obliterans (Vascular disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis infective (Infections and infestations) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 4 | 4
Cardiac death (General disorders) | 1 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 3
Carotid artery disease (Nervous system disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 4
Cellulitis (Infections and infestations) | 4 | 6
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 5 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Discomfort (General disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Epilepsy (Nervous system disorders) | 0 | 1
Gangrene (Infections and infestations) | 1 | 4
Generalised oedema (General disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 3
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 2 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 3 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 1
Periproctitis (Gastrointestinal disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Postoperative wound infection (Infections and infestations) | 2 | 5
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 17 | 10
Respiratory tract infection (Infections and infestations) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Skin injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 3 | 2
Subileus (Gastrointestinal disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Tremor (Nervous system disorders) | 1 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urinary tract infection (Infections and infestations) | 8 | 9
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Ventricular asystole (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 8 | 11
Accelerated hypertension (Vascular disorders) | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Anal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 3 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2
Bacteraemia (Infections and infestations) | 1 | 1
Basilar migraine (Nervous system disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 3
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Coronary artery insufficiency (Cardiac disorders) | 1 | 1
Coronary artery occlusion (Cardiac disorders) | 3 | 4
Coronary artery stenosis (Cardiac disorders) | 20 | 16
Diverticulitis (Infections and infestations) | 0 | 1
Drug withdrawal syndrome (General disorders) | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 69 | 23
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypertensive crisis (Vascular disorders) | 5 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 8
Hypotension (Vascular disorders) | 5 | 3
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 3
Ischaemic gastritis (Gastrointestinal disorders) | 0 | 1
Ischaemic ulcer (General disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 3
Leriche syndrome (Vascular disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Nephrolithiasis (Renal and urinary disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 38 | 46
Pharyngoesophageal diverticulum (Gastrointestinal disorders) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 5 | 7
Silicosis (Injury, poisoning and procedural complications) | 0 | 1
Spinal cord haemorrhage (Nervous system disorders) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 4
Arterial thrombosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 2 | 0
Artery dissection (Vascular disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 1
Bladder diverticulum (Renal and urinary disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 94 | 82
Cardio-respiratory arrest (Cardiac disorders) | 1 | 3
Chronic sinusitis (Infections and infestations) | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Dressler's syndrome (Cardiac disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 2 | 0
Endocarditis (Infections and infestations) | 1 | 2
Eye haemorrhage (Eye disorders) | 2 | 0
Fatigue (General disorders) | 0 | 1
Femoral arterial stenosis (Vascular disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 4 | 2
Gastritis erosive (Gastrointestinal disorders) | 1 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 2
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 4
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 2 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Maculopathy (Eye disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Renal injury (Renal and urinary disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 2 | 2
Rib fracture (Injury, poisoning and procedural complications) | 0 | 4
Sick sinus syndrome (Cardiac disorders) | 0 | 3
Sinus bradycardia (Cardiac disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 2
Anaemia (Blood and lymphatic system disorders) | 16 | 8
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 2 | 0
Appendicitis (Infections and infestations) | 4 | 0
Arrhythmia (Cardiac disorders) | 4 | 1
Arterial stenosis (Vascular disorders) | 1 | 0
Asthenia (General disorders) | 0 | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 5
Biliary colic (Hepatobiliary disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 2 | 7
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 2 | 0
Epiglottitis (Infections and infestations) | 0 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Fat embolism (Injury, poisoning and procedural complications) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 12 | 6
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 5 | 4
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Intermittent claudication (Vascular disorders) | 1 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Laryngeal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Peripheral embolism (Vascular disorders) | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Rectal fissure (Gastrointestinal disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 8 | 5
Renal infarct (Renal and urinary disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Septic shock (Infections and infestations) | 4 | 2
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Spinal cord ischaemia (Nervous system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 2 | 0
Ventricular fibrillation (Cardiac disorders) | 8 | 5
Wound infection (Infections and infestations) | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 26 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac perforation (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 5 | 2
Clostridium test positive (Investigations) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 1 | 0
Death (General disorders) | 11 | 8
Device dislocation (General disorders) | 1 | 3
Device related sepsis (Infections and infestations) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 4 | 2
Diverticulum (Gastrointestinal disorders) | 2 | 1
Dizziness (Nervous system disorders) | 4 | 6
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Encephalitis herpes (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 2 | 2
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 5
Gastrointestinal infection (Infections and infestations) | 2 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Haematuria (Renal and urinary disorders) | 13 | 5
Haemoglobin decreased (Investigations) | 4 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 2
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Injection site infection (Infections and infestations) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Ischaemia (Vascular disorders) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Laryngitis (Infections and infestations) | 0 | 2
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 150 | 158
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 2
Occult blood positive (Investigations) | 2 | 0
Parasystole (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Presyncope (Nervous system disorders) | 2 | 3
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Testis cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Ventricle rupture (Cardiac disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 5 | 2
Acute prerenal failure (Renal and urinary disorders) | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Angina unstable (Cardiac disorders) | 157 | 157
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchitis (Infections and infestations) | 6 | 1
Bronchopneumonia (Infections and infestations) | 0 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Chest pain (General disorders) | 11 | 7
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 14 | 8
Completed suicide (Psychiatric disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 6 | 3
Coronary artery dissection (Cardiac disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 1
Depression (Psychiatric disorders) | 0 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Femoral artery aneurysm (Vascular disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Gallbladder empyema (Infections and infestations) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Haematocrit decreased (Investigations) | 1 | 0
Haematoma (Vascular disorders) | 14 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemorrhage (Vascular disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 8 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 4 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Pain (General disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Panic disorder (Psychiatric disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 4 | 0
Pericardial haemorrhage (Cardiac disorders) | 3 | 4
Periodontitis (Gastrointestinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 1
Pyrexia (General disorders) | 3 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Renal impairment (Renal and urinary disorders) | 5 | 6
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 2 | 0
Sudden cardiac death (General disorders) | 10 | 11
Syncope (Nervous system disorders) | 13 | 14
Tracheobronchitis (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 3 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 3 | 1
Ventricular arrhythmia (Cardiac disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Wound (Injury, poisoning and procedural complications) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 2 | 0
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 6 | 3
Bacterial sepsis (Infections and infestations) | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0
Bladder cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Bradycardia (Cardiac disorders) | 9 | 3
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1
Carotid arteriosclerosis (Nervous system disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 6 | 3
Cholestasis (Hepatobiliary disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Convulsion (Nervous system disorders) | 2 | 0
Coronary artery disease (Cardiac disorders) | 22 | 18
Dehydration (Metabolism and nutrition disorders) | 4 | 4
Dementia (Nervous system disorders) | 1 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 2
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Drug screen positive (Investigations) | 1 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Fungal skin infection (Infections and infestations) | 1 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Hypertensive emergency (Vascular disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 0
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 7 | 7
Infected bites (Infections and infestations) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 2 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 2
Intraventricular haemorrhage (Nervous system disorders) | 5 | 0
Left ventricular dysfunction (Cardiac disorders) | 2 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mental retardation (Nervous system disorders) | 0 | 1
Multi-organ failure (General disorders) | 4 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Myocardial rupture (Cardiac disorders) | 1 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nephropathy (Renal and urinary disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 3 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Paraplegia (Nervous system disorders) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 4 | 4
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 3 | 2
Sciatica (Nervous system disorders) | 2 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 2
Subcutaneous abscess (Infections and infestations) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban 5 mg BID (N=3672) | Placebo BID (N=3643)
Chest pain (General disorders) | 186 | 173
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 186 | 63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.